CLINICAL TRIAL: NCT02058433
Title: Phase 3, Randomized, Open-label Study of the Safety of Individual Paclitaxel Dose Adjustment Based on Pharmacokinetic Follow up Versus Conventional Dosage in First-line Treatment in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety Study of Individual Paclitaxel Dose Adjustment Based on Pharmacokinetics in Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caicun Zhou (Other)
Responsible Party: Sponsor-Investigator, Caicun Zhou, Tonji University Affiliated Shanghai Pulmonary Hospital, Tongji University
Organization: Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPAP
Record Dates: First submitted 2014-01-27; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Chemotherapy; Individual Paclitaxel dose; pharmacokinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pharmacokinetics group (Experimental): Based on pharmacokinetics. Observe safety and efficacy. In first cycle a fixed Paclitaxel dose depends on BSA. In subsequent cycles the dosage of Paclitaxel will be adjusted depending on pharmacokinetics follow up .
  Interventions: Other: dosage of paclitaxel
- Body surface area(BSA) group (Active Comparator): Based on body surface area. The dosage of Paclitaxel is based on the BSA of the patient. Paclitaxel/carboplatin up to 4 cycles or disease progression or intolerable toxicity.
  Interventions: Other: dosage of paclitaxel

INTERVENTIONS:
Other: dosage of paclitaxel — Based on pharmacokinetics. Observe the toxicity in an individual patient after a fixed Paclitaxel dose depending on BSA and then the dosage of Paclitaxel is adjusted depending on pharmacokinetics follow up to avoid excess toxicity in subsequent cycles.
  Arms: pharmacokinetics group
Other: dosage of paclitaxel — Based on body surface area. The dosage of Paclitaxel is based on the BSA of the patient. Paclitaxel/carboplatin up to 4 cycles or disease progression or intolerable toxicity.
  Arms: Body surface area(BSA) group

SUMMARY:
Platinum-based doublets including paclitaxel, gemcitabine, or docetaxel are standard 1st regimens in Non-Small Cell Lung Cancer(NSCLC). The traditional method of individualizing cytotoxic drug dose is by using body surface area(BSA), which is not correlated with the ability of an individual to metabolize or excrete cytotoxic drugs, because it is not related to liver function and is poorly correlated with glomerular filtration rate, and does not seem to be a determinant of toxicity. Pharmacokinetic parameters such as area under the curve have been shown to correlate with toxicity. The advantages of using a fixed dose of antineoplastic agents for all of the patients are obvious. Pharmacokinetically guided treatment would avoid severe adverse effects, which has not been sufficiently investigated in advanced NSCLC.First, the investigators monitor the blood concentrations of paclitaxel and neutropenia blood toxicity after chemotherapy with paclitaxel and carboplatin in patients of NSCLC and verify suitable paclitaxel therapeutic window for Chinese patients. Then the investigators compare safety and efficacy between individual paclitaxel dose adjustment based on the therapeutic window compared with conventional dosage.

DETAILED DESCRIPTION:
Primary end point: Common Terminology Criteria for Adverse Events(CTCAE) grade 4.

Secondary end point:Objective Response Rate(ORR),Progression Free Survival(PFS),Overall Survival(OS),Quality Of Life(QOL) etc.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study treatment period patients must fulfil all of the following criteria:

1. Provision of informed consent.
2. Male or female aged 18 years and over.
3. Histologically or cytologically confirmed non-small cell lung carcinoma.
4. Locally advanced Stage not amenable to local therapy (e.g. pleural effusion) or metastatic disease.
5. No prior chemotherapy, biological (including targeted therapies such as Epidermal Growth Factor Receptor(EGFR) and Vascular Epidermal Growth Factor (VEGF) inhibitors) or immunological therapy. Patients who are willing to accept with paclitaxel and carboplatin as adjuvant chemotherapy will be eligible.
6. World Health Organization (WHO) performance status (PS) of 0 to 2.
7. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.
8. Laboratory values within the range, as defined below, within two weeks of randomization:

   * Absolute neutrophils count(ANC)≥2.0×109/L
   * Platelets≥100×109/L
   * Serum bilirubin≤2×ULN; Aspartate transaminase(AST) and alanine tansaminase (ALT) ≤2.5×ULN(≤5×ULN if liver metastases)
   * Creatinine clearance≥60ml/min
9. Measurable disease according to Response Evaluation Criteria in Solid Tumors(RECIST) criteria with at least one measurable lesion not previously irradiated.
10. Life expectancy ≥12 weeks.

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
2. Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
3. Known severe hypersensitivity to carboplatin, paclitaxel or any of the excipients of these products.Known severe hypersensitivity to pre-medications required for treatment with carboplatin / paclitaxel doublet chemotherapy.
4. Prior treatment with paclitaxel.
5. Current treatment with target drug and biological therapy.
6. Pregnant or lactating woman.
7. Prior chemotherapy, biological (including targeted therapies such as Epidermal Growth Factor Receptor(EGFR) and Vascular Epidermal Growth Factor (VEGF) inhibitors) or immunological therapy were received even if treatment was not paclitaxel and was completed in 4 weeks before day1 of study treatment.
8. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
9. Life expectancy of less than 12 weeks.
10. Unable to tolerate carboplatin / paclitaxel doublet chemotherapy, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
CTCAE grade 4 of the blood marrow | 24 months
  Record the number of CTCAE grade 4 of the blood marrow such as Leukocytes, Neutrophils,Platelets and Hemoglobin in two treatment groups since the initiation of chemotherapy

SECONDARY OUTCOMES:
Objective response rate | Tumor assessment 6-8 weeks after the initiation of chemotherapy
  The objective tumour response rate will be calculated as the percentage of evaluable patients with complete response (CR) and partial response (PR).
Progression free survival | 12 months
  Progression Free Survival (PFS) is defined as the time from randomization to the first documentation of objective disease progression (PD) or death from any cause.
Overall survival | 24 months
  Overall survival(OS) is defined as the interval between the date of randomization and the date of patient death due to any cause, or the last date the patient was known to be alive.
Quality of life | 24 months
  Data on QoL will be assessed using the Functional Assessment of Cancer Therapy - Lung (FACT-L) for every patients.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Ph.D, Principal Investigator — Tongji University Affiliated Shanghai Pulmonary Hospital
Locations (1):
- Medical Department, Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Zhou F, Qi H, Ni H, Hu Q, Zhou C, Li Y, Baburina I, Courtney J, Salamone SJ. Randomized study of individualized pharmacokinetically-guided dosing of paclitaxel compared with body-surface area dosing in Chinese patients with advanced non-small cell lung cancer. Br J Clin Pharmacol. 2019 Oct;85(10):2292-2301. doi: 10.1111/bcp.13982. Epub 2019 Jun 14. PMID 31077432